CLINICAL TRIAL: NCT06274723
Title: Identifying and Examining the Effects of Source and Presentation on Responses to Electronic Cigarette Public Education Messages in Young Adult Vapers and Non-vapers - Part 1
Brief Title: Responses to E-cigarette Message Source and Presentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Donghee Nicole Lee, Postdoctoral Fellow, University of Massachusetts, Worcester
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00001220; 1K99CA281094-01A1 (NIH)
Record Dates: First submitted 2024-01-17; First posted 2024-02-23 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Vaping
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Expert, one-sided (Experimental): Participants assigned to the expert, one-sidedness condition will receive one-sided e-cigarette messages from an expert source.
  Interventions: Other: Expert, one-sided
- Expert, two-sided (Experimental): Participants assigned to the expert, two-sidedness condition will receive two-sided e-cigarette messages from an expert source.
  Interventions: Other: Expert, two-sided
- Peer, one-sided (Experimental): Participants assigned to the peer, one-sidedness condition will receive one-sided e-cigarette messages from a peer source.
  Interventions: Other: Peer, one-sided
- Peer, two-sided (Experimental): Participants assigned to the peer, two-sidedness condition will receive two-sided e-cigarette messages from a peer source.
  Interventions: Other: Peer, two-sided

INTERVENTIONS:
Other: Expert, one-sided — Participants will view a brief description of an expert source and see one-sided e-cigarette education messages.
  Arms: Expert, one-sided
Other: Expert, two-sided — Participants will view a brief description of an expert source and see two-sided e-cigarette education messages.
  Arms: Expert, two-sided
Other: Peer, one-sided — Participants will view a brief description of a peer source and see one-sided e-cigarette education messages.
  Arms: Peer, one-sided
Other: Peer, two-sided — Participants will view a brief description of a peer source and see two-sided e-cigarette education messages.
  Arms: Peer, two-sided

SUMMARY:
The goal of this clinical trial is to use crowdsourcing to test the effects of a message source (expert and peer) and message presentation types (one-sided and two-sided) to identify the optimal message type for young adults who vape and do not vape.

ELIGIBILITY:
Inclusion Criteria:

* US residents ages 18-24
* Fluent in English
* Reporting either vaping in the past 30 days or not having vaped in the past 30 days but susceptible to vaping

Exclusion Criteria:

* Age less than 18 or above 24
* Not fluent in English
* Not a member of partnering crowdsourcing behavioral research platform conducting the study

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 848 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donghee N Lee, PhD, Principal Investigator — UMass Chan Medical School
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: n=109 data were removed from analysis; if 1) study duration was less than the average study duration (i.e., 8 minutes; n=44, if the participant age exceeded the eligible age (n=19); and if non-vapers did not meet the susceptibility criteria (n=46).
Groups:
- Expert, One-Sided: Participants assigned to the expert, one-sidedness condition were first presented with a brief description of a expert source. They then viewed an e-cigarette message that discussed only the health harms of e-cigarette use. This sequence was repeated 18 times during a single study visit.
- Expert, Two-Sided: Participants assigned to the expert, two-sidedness condition were first presented with a brief description of an expert source. They then viewed an e-cigarette message that acknowledged both the potential benefits of e-cigarette use and the associated health risks. This sequence was repeated 18 times during a single study visit.
- Peer, One-Sided: Participants assigned to the peer, one-sidedness condition were first presented with a brief description of a peer source. They then viewed an e-cigarette message that discussed only the health harms of e-cigarette use. This sequence was repeated 18 times during a single study visit.
- Peer, Two-Sided: Participants assigned to the peer, two-sidedness condition were first presented with a brief description of an peer source. They then viewed an e-cigarette message that acknowledged both the potential benefits of e-cigarette use and the associated health risks. This sequence was repeated 18 times during a single study visit.
Period: Overall Study
Arm/Group | Expert, One-Sided | Expert, Two-Sided | Peer, One-Sided | Peer, Two-Sided
Started | 209 | 208 | 210 | 210
Completed | 191 | 197 | 203 | 194
Not Completed | 18 | 11 | 7 | 16

BASELINE CHARACTERISTICS:
Groups:
- Expert, One-Sided: Participants first saw a brief description of a expert source. Then they viewed an e-cigarette message that discussed only the health harms of e-cigarette use. This sequence was repeated 18 times during a single study visit.
- Expert, Two-Sided: Participants first saw a brief description of an expert source. They then viewed an e-cigarette message that acknowledged both the potential benefits of e-cigarette use and the associated health risks. This sequence was repeated 18 times during a single study visit.
- Peer, One-Sided: Participants first saw a brief description of a peer source. They then viewed an e-cigarette message that discussed only the health harms of e-cigarette use. This sequence was repeated 18 times during a single study visit.
- Peer, Two-Sided: Participants first saw a brief description of an peer source. They then viewed an e-cigarette message that acknowledged both the potential benefits of e-cigarette use and the associated health risks. This sequence was repeated 18 times during a single study visit.
- Total: Total of all reporting groups
Arm/Group | Expert, One-Sided | Expert, Two-Sided | Peer, One-Sided | Peer, Two-Sided | Total
Number analyzed (Participants) | 191 | 197 | 203 | 194 | 785
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.04 (1.79) | 21.78 (1.77) | 21.88 (1.69) | 21.85 (1.83) | 21.89 (1.77)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 89 | 101 | 92 | 88 | 370
  Male | 93 | 83 | 101 | 92 | 369
  Others | 9 | 13 | 10 | 14 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 24 | 29 | 26 | 102
  Not Hispanic or Latino | 168 | 173 | 174 | 168 | 683
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 2 | 5
  Asian | 21 | 20 | 18 | 22 | 81
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 1 | 3
  Black or African American | 43 | 50 | 49 | 53 | 195
  White | 97 | 96 | 98 | 88 | 379
  More than one race | 10 | 16 | 8 | 13 | 47
  Unknown or Not Reported | 18 | 15 | 27 | 15 | 75
Region of Enrollment [Number; unit: participants]
  United States | 191 | 197 | 203 | 194 | 785
Vaping status [Count of Participants; unit: Participants]
  Current vapers | 103 | 112 | 115 | 100 | 430
  Susceptible non-vapers | 79 | 74 | 74 | 82 | 309
  Others | 9 | 11 | 14 | 12 | 46

OUTCOME MEASURES:

1. Primary Outcome: Message Acceptance
Description: Participants' self-reported message acceptance were measured by using a five-point Likert scale using five items assessing whether participants thought the message was worth remembering, grabbed their attention, powerful, convincing, and meaningful on a scale from 1 (Strongly disagree) to 5 (Strongly agree). Items were summed and averaged to create a single composite score, and this was done for each arm for each vaping status. Higher scores indicate more more message acceptance, therefore better outcomes.
Time Frame: After exposure to each messages (approximately up to 20 minutes total), measured during a single study visit on Day 1.
Population: The data were stratified based on participants' vaping status ("Current vapers" and "Susceptible non-vapers"). The Number of Participants Analyzed for each row reflects the actual number of participants within that vaping status group who were included in the analysis. The Overall Number of Participants Analyzed represents the total number of both subgroups. Any differences have been clarified to specify participant numbers at the row level.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Expert, One-Sided | Expert, Two-Sided | Peer, One-Sided | Peer, Two-Sided
Number analyzed (Participants) | 182 | 186 | 189 | 182
units on a scale
  Current vapers: number analyzed (Participants) | 103 | 112 | 115 | 100
  Current vapers | 3.01 (0.01) | 3.00 (0.01) | 2.88 (0.01) | 2.76 (0.01)
  Susceptible non-vapers: number analyzed (Participants) | 79 | 74 | 74 | 82
  Susceptible non-vapers | 2.94 (0.09) | 2.77 (0.03) | 2.77 (0.09) | 2.72 (0.09)

2. Primary Outcome: Harm Perceptions
Description: Harm perceptions was measured by a single item e-cigarette harm perceptions question assessing participants' perceived absolute harm of e-cigarette use on a scale from 1 (Not at all harmful) to 10 (Very harmful). Items were summed and averaged to create a single composite score. This was done for each vaping status (current vapers and susceptible non-vapers). Higher scores indicate greater vaping harm perceptions, therefore indicating better outcome.
Time Frame: After exposure to each messages (approximately up to 20 minutes total), measured during a single study visit on Day 1.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Expert, One-Sided | Expert, Two-Sided | Peer, One-Sided | Peer, Two-Sided
Number analyzed (Participants) | 182 | 186 | 189 | 182
units on a scale
  Current vapers: number analyzed (Participants) | 103 | 112 | 115 | 100
  Current vapers | 7.39 (0.20) | 7.45 (0.19) | 7.27 (0.19) | 7.44 (0.20)
  Susceptible non-vapers: number analyzed (Participants) | 79 | 74 | 74 | 82
  Susceptible non-vapers | 8.05 (0.19) | 8.04 (0.20) | 8.04 (0.20) | 7.82 (0.19)

3. Secondary Outcome: Negative Cognition
Description: Negative cognition was measured by six-item reactance questionnaire, such as perceptions of messages being manipulative, misleading, distorted, overblown, exaggerated, and overstated on a scale from 1 (Strongly disagree) to 5 (Strongly agree). Higher scores indicate greater negative cognition, indicating worse outcome.
Time Frame: After exposure to each messages (approximately up to 20 minutes total), measured during a single study visit on Day 1.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Expert, One-Sided | Expert, Two-Sided | Peer, One-Sided | Peer, Two-Sided
Number analyzed (Participants) | 182 | 186 | 189 | 182
units on a scale
  Current vapers: number analyzed (Participants) | 103 | 112 | 115 | 100
  Current vapers | 3.79 (0.08) | 3.81 (0.08) | 3.87 (0.08) | 3.78 (0.08)
  Susceptible non-vapers: number analyzed (Participants) | 79 | 74 | 74 | 82
  Susceptible non-vapers | 4.00 (0.08) | 4.17 (0.09) | 4.12 (0.09) | 4.12 (0.08)

4. Secondary Outcome: Message Anger
Description: Message anger was measured by four item message anger question assessing the extent to which the messages made participants feel irritated, angry, annoyed, and aggravated on a scale from 1 (not at all) to 5 (very much). Items were summed and averaged. This was done for each vaping status (current vapers and susceptible non-vapers). Higher scores indicate greater anger toward messages, indicating worse outcomes.
Time Frame: After exposure to each messages (approximately up to 20 minutes total), measured during a single study visit on Day 1.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Expert, One-Sided | Expert, Two-Sided | Peer, One-Sided | Peer, Two-Sided
Number analyzed (Participants) | 182 | 186 | 189 | 182
units on a scale
  Current vapers: number analyzed (Participants) | 103 | 112 | 115 | 100
  Current vapers | 4.07 (0.08) | 4.12 (0.08) | 4.19 (0.08) | 4.05 (0.08)
  Susceptible non-vapers: number analyzed (Participants) | 79 | 74 | 74 | 82
  Susceptible non-vapers | 4.42 (0.07) | 4.57 (0.07) | 4.54 (0.07) | 4.56 (0.07)

5. Secondary Outcome: Message Liking
Description: Message liking will be measured by a single-item liking of the message on scale from 1 (Dislike very much) to 5 (Like very much). Items were summed and averaged to create a single composite score. This was done for each vaping status (current vapers and susceptible non-vapers). Higher scores indicate greater message liking, therefore indicating better outcome.
Time Frame: After exposure to each messages (approximately up to 20 minutes total), measured during a single study visit on Day 1.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Expert, One-Sided | Expert, Two-Sided | Peer, One-Sided | Peer, Two-Sided
Number analyzed (Participants) | 182 | 186 | 189 | 182
units on a scale
  Current vapers: number analyzed (Participants) | 103 | 112 | 115 | 100
  Current vapers | 3.08 (0.09) | 3.05 (0.08) | 2.95 (0.08) | 2.97 (0.09)
  Susceptible non-vapers: number analyzed (Participants) | 79 | 74 | 74 | 82
  Susceptible non-vapers | 3.03 (0.07) | 2.97 (0.07) | 3.02 (0.07) | 3.00 (0.07)

6. Secondary Outcome: Source Trust
Description: Source trust was measured by a single-item trust in health information source questionnaire, such as trust in source about vaping information on a scale from 1(Not at all) to 5 (Very much so). Items were summed and averaged to create a single composite score. This was done for each vaping status (current vapers and susceptible non-vapers). Higher scores indicate greater source trust, therefore indicating better outcome
Time Frame: After exposure to each messages (approximately up to 20 minutes total), measured during a single study visit on Day 1.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Expert, One-Sided | Expert, Two-Sided | Peer, One-Sided | Peer, Two-Sided
Number analyzed (Participants) | 182 | 186 | 189 | 182
units on a scale
  Current vapers: number analyzed (Participants) | 103 | 112 | 115 | 100
  Current vapers | 3.13 (0.09) | 3.21 (0.08) | 2.99 (0.08) | 3.01 (0.09)
  Susceptible non-vapers: number analyzed (Participants) | 79 | 74 | 74 | 82
  Susceptible non-vapers | 3.27 (0.08) | 3.32 (0.08) | 3.01 (0.08) | 2.96 (0.08)

7. Secondary Outcome: Attitudes
Description: Participants' self-reported vaping attitudes were measured by using a five-point bipolar scale using 7 subscale items assessing whether participants thought vaping was enjoyable, healthy, safe, fun, smart, cool, and attractive on a scale from 1 (negative attitudes) to 5 (positive attitudes). Items were summed and averaged to create a single composite score, and this was done for each arm for each vaping status. Higher scores indicate more positive e-cigarette attitudes, therefore worse outcomes.
Time Frame: After exposure to all messages (approximately up to 45 minutes), measured during a single study visit on Day 1.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Expert, One-Sided | Expert, Two-Sided | Peer, One-Sided | Peer, Two-Sided
Number analyzed (Participants) | 182 | 186 | 189 | 182
units on a scale
  Current vapers: number analyzed (Participants) | 103 | 112 | 115 | 100
  Current vapers | 2.57 (0.76) | 2.66 (0.81) | 2.73 (0.83) | 2.61 (0.8)
  Susceptible non-vapers: number analyzed (Participants) | 79 | 74 | 74 | 82
  Susceptible non-vapers | 1.51 (0.81) | 1.53 (0.94) | 1.41 (0.72) | 1.33 (0.59)

8. Secondary Outcome: Behavioral Intentions to Vape or Try Vaping
Description: Participants' vaping or vaping trial intentions were measured by using a 3 subscale items assessing participants' intentions to vape: soon/anytime during the next year/would use offered by one of their best friends, on a scale from 1 (Definitely not) to 5 (Definitely yes). Items were summed and averaged to create a single composite score. This was done for each vaping status (current vapers and susceptible non-vapers). Higher scores indicate greater vaping intentions, therefore indicating worse outcome.
Time Frame: After exposure to all messages (approximately up to 45 minutes), measured during a single study visit on Day 1.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Expert, One-Sided | Expert, Two-Sided | Peer, One-Sided | Peer, Two-Sided
Number analyzed (Participants) | 182 | 186 | 189 | 182
units on a scale
  Current vapers: number analyzed (Participants) | 103 | 112 | 115 | 100
  Current vapers | 3.08 (1.1) | 2.88 (1.14) | 3.05 (1.23) | 3.07 (1.15)
  Susceptible non-vapers: number analyzed (Participants) | 79 | 74 | 74 | 82
  Susceptible non-vapers | 1.51 (0.81) | 1.53 (0.94) | 1.41 (0.72) | 1.33 (0.59)

ADVERSE EVENTS:
Time Frame: Each adverse event or serious adverse event was monitored and assessed throughout the entire duration of the participant's study participation, from the moment a participant clicked on the study link until the study completed, which lasted approximately 45 minutes per participant during a single study visit on Day 1.
Description: The study used a non-systematic assessment method, where adverse events were monitored through participants' reports (direct message to the research team via the crowdsourcing website). No adverse events were reported by participants or observed during the study duration.
Arm/Group | Expert, One-sided | Expert, Two-sided | Peer, One-sided | Peer, Two-sided
All-Cause Mortality (participants affected / at risk) | 0/191 | 0/197 | 0/203 | 0/194
Serious Adverse Events (participants affected / at risk) | 0/191 | 0/197 | 0/203 | 0/194
Other Adverse Events (participants affected / at risk) | 0/191 | 0/197 | 0/203 | 0/194

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT06274723/Prot_001.pdf
  • Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT06274723/SAP_000.pdf